CLINICAL TRIAL: NCT05180318
Title: Effects of Esketamine Pre-administration on Blood Lymphocyte Subsets and Inflammatory Factors in Early Postoperative Period:
Brief Title: Prophylactic Effects of Esketamine in Surgical Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiancheng Zhang, Principal investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WJ-2020-01
Record Dates: First submitted 2021-12-01; First posted 2022-01-06 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Surgical Injury
Keywords: Esketamine; Inflammatory cytokines; Lymphocyte subsets
MeSH Terms: conditions — Intraoperative Complications | interventions — Esketamine; Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.9% saline preadministration group (Placebo Comparator): 0.9% saline will be given intravenously 24-36 hours before operation and immediately after operation
  Interventions: Drug: 0.9% saline
- Esketamine preadministration group (Experimental): Esketamine (0.25 mg/kg) will be given intravenously 24-36 hours before surgery (infusion time: 40 min) and immediately after surgery (infusion time: 40 min).
  Interventions: Drug: Esketamine Hydrochloride 28 Mg in 0.2 mL NASAL SOLUTION [Spravato]

INTERVENTIONS:
Drug: Esketamine Hydrochloride 28 Mg in 0.2 mL NASAL SOLUTION [Spravato] — Esketamine (0.25 mg/kg) will be given intravenously 24-36 hours before surgery (infusion time: 40 min) and immediately after surgery (infusion time: 40 min).
  Other Names: (S)-ketamine
  Arms: Esketamine preadministration group
Drug: 0.9% saline — 0.9% saline
  Arms: 0.9% saline preadministration group

SUMMARY:
Evidences have showing that esketamine has anti-inflammatory and therapeutic effects on depression and cardiac surgery. The investigators' preliminary results suggest that combined prophylactic and therapeutic use of esketamine could decrease the plasma levels of pro-inflammatory cytokines after LPS-induced endotoxemia. The investigators also found that combined prophylactic and therapeutic use of esketamine could attenuate systemic inflammation and inflammatory multi-organ injury in mice after CLP-induced lethal sepsis.

Surgical trauma could elicit a marked inflammatory response with increased expression of pro-inflammatory cytokines, as well as postoperative immunosuppression. However, it remains unclear whether combined prophylactic and therapeutic use of esketamine could improve postoperative immunosuppression and alleviates systemic inflammatory response.

This project aims to study whether combined prophylactic and therapeutic use of esketamine could improve the decreased number of lymphocyte subsets and increased plasma pro-inflammatory cytokines.

DETAILED DESCRIPTION:
Esketamine is a new antidepressant approved by the US Food and Drug Administration (FDA) in 2019. It has rapid action and accurate treatment effect for refractory severe depression. Studies have shown that esketamine also has significant anti-inflammatory effects. The investigators' previous study found that esketamine has a good preventive effect on inflammatory response, but the effect of preoperative preadministration of esketamine on postoperative systemic immune function and systemic inflammatory response is not clear.

Clinical studies have shown that esketamine (0.25 mg/kg, 40 min infusion time) can rapidly improve the depressive symptoms of patients with treatment-resistant depression. Esketamine is shown to be able to play a neuroprotective role by reducing glial cell activation and the production of inflammatory cytokines such as tumor necrosis factor (TNF-α) and interleukin-6 (IL-6). Esketamine at a dose of 0.2 mg/kg or 0.4 mg/kg has significant antidepressant effects in the treatment of resistant depression. The antidepressant effects of esketamine may be closely related to its anti-inflammatory effect. During cardiopulmonary bypass surgery, anesthesia induction was supplemented with 1-3 mg/kg esketamine, anesthesia maintenance was supplemented with 2-3 mg/kg/h esketamine, anesthesia maintenance time was 283 minutes, the total amount of esketamine was 1580mg on average. Esketamine decreased plasma levels of IL-6 (6 h after opening the aorta) and IL-8 (1 and 6 h after opening the aorta) and increased plasma levels of IL-10 (1 h after opening the aorta). In the investigators' preliminary study on the role of esketamine in systemic inflammation induced by lipopolysaccharide (LPS), the investigators found that in systemic LPS (5 mg/kg)-induced systemic inflammation model, esketamine (10 mg/kg, IP) was administrated twice 24 hours before LPS administration and 10 minutes after LPS administration. The plasma levels of IL-6, IL-17A and interferon γ (IFN-γ) were significantly decreased 24 h after LPS administration in mice. Single administration of esketamine 10 min after LPS administration did not significantly reduce the plasma levels of IL-6 and IL-17A at 24 h. The investigators further found that in mice with LPS (8 mg/kg)-induced systemic inflammation, twice intraperitoneal administration of esketamine (10 mg/kg, IP) 24 hours before LPS administration and 10 minutes after LPS administration also significantly reduced the plasma levels of IL-17A 24 hours after LPS administration. Surgery-induced trauma could cause significant inflammatory responses, manifested by increased expression of pro-inflammatory cytokines. Studies have found that ketamine at a dose of 0.5 mg/kg administrated immediately before chest surgery could reduce the plasma levels of IL-6 and C-reactive protein 24 hours after surgery. However, it remains unclear whether preoperative and immediate postoperative administration of esketamine could improve postoperative immune function and alleviate systemic inflammatory response.

The investigators will include patients subjected to elective surgery strictly according to the inclusion and exclusion criteria to investigate whether preoperative and immediate postoperative administration of esketamine has postoperative anti-inflammatory effects on postoperative delirium, postoperative pain, and postoperative sleep, as well as on total length of hospital stay, in-hospital infection complications, in-hospital mortality, and 90-day readmission rates. Prophylactic administration of esketamine before surgery is expected to provide a new therapeutic strategy for alleviating postoperative systemic inflammation and improving postoperative immune suppression.

Enrolled patients were randomly assigned to two groups: the esketamine preadministration group and the placebo control group. Esketamine at a dose of 0.25 mg/kg (40 min infusion time) or normal saline was given intravenously 24-36 hours before surgery, and esketamine at a dose of 0.25 mg/kg (40 min infusion time) or normal saline was given intravenously immediately after surgery.

Seven tubes of venous blood were collected and sent to the laboratory and immunology department of Union Hospital affiliated to Tongji Medical College, Huazhong University of Science and Technology, 24 hours before and after the first administration of esketamine, and seven tests including blood routine, coagulation, liver function, kidney function, electrolytes, C-reactive protein, myocardial enzyme, BNP, lymphocyte subsets and cytokines were performed. A tube of venous blood was taken at each of the two time points in the study and centrifuged to obtain plasma, which was frozen and stored at -80℃ for ELISA detection of ANP.

If the adverse events of esketamine appear during the study, patients or authorized client withdraw from the study actively, or drugs that seriously affect systemic inflammation and immune function (such as non-steroidal anti-inflammatory drugs, immunosuppressants, immunoenhancers, high doses of hormones (more than 10mg prednisolone per day or equivalent dose of other hormones, etc.) were used in clinical treatment, the study will be terminated. In this study, adverse reactions were evaluated daily and closely monitored within 7 days after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old without restriction of gender, race, religion, creed or nationality;
* Surgery with general anesthesia operation with estimated operation time of at least 2 hours;
* Patients and/or their family members know and agree to participate in the trial.

Exclusion Criteria:

* Local anesthesia surgery;
* Being admitted to ICU immediately after surgery;
* Pregnant or breastfeeding;
* History of solid organ or bone marrow transplantation;
* Diseases that may affect immune-related indicators, including autoimmune diseases (rheumatoid arthritis and systemic lupus erythematosus, etc.), and malignant hematological tumours (leukaemia and lymphoma, etc.);
* Acute brain injury, including traumatic brain injury, subarachnoid hemorrhage, acute ischemic stroke, acute intracranial hemorrhage and acute intracranial infection;
* Chronic nephrosis;
* Acute myocardial infarction or severe heart failure (NYHA: Grade 4);
* Severe chronic liver disease (child-Pugh: Grade C);
* Deafness, aphasia, mental illness or severe cognitive impairment;
* Endotracheal intubation could not be removed within 24 hours after surgery
* Patients and/or their family members refuse to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery percentage of peripheral blood lymphocyte subsets | 24 hours after surgery
  CD3+、CD3+CD4+、CD3+CD8+、CD3-CD16+CD56+ NK cells、CD19+ B cells
Deterioration percentage of peripheral blood pro-inflammatory cytokines | 24 hours after surgery
  IL-2、IL-4、IL-6、IL-10、IL-17A、IFN-γ、TNF-α

SECONDARY OUTCOMES:
Plasma levels of atrial natriuretic peptide (ANP) | At 24 hours after surgery
  The protein expression of ANP in the plasma.
Recovery percentage of peripheral blood neutrophil to lymphocyte ratio (NLR) | At 24 hours after surgery
  [NLR (24 hours)-NLR (baseline)]/NLR (baseline)×100%
Total length of hospital stay | Up to 24 weeks
  The time from admission to discharge.
Infectious complications after inclusion during hospitalization | Up to 24 weeks
  Lung infection, bloodstream infection and surgical wound infection, etc.
28-day mortality rate | Up to 28 days after inclusion
  Death within 28 days after hospitalization.
90-day readmission rate | Up to 90 days after discharge from hospital
  Hospitalized again within 90 days after discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jiancheng Zhang, MD, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
After publication, the data supporting the findings of this study can be provided by the corresponding author upon reasonable request. Participant data without names and identifiers can be provided by the corresponding author and the Wuhan Union Hospital after approval. The research team will provide an email address for communication purposes once approval is obtained regarding sharing the data with others. The proposal with detailed description of the study objectives and statistical analysis plan will be needed for evaluation of the purpose for the data request. Additional materials may also be required during the process of evaluation.
Supporting Information: Study Protocol
Time Frame: Six months after publication.
Access Criteria: Upon reasonable request.